CLINICAL TRIAL: NCT05934552
Title: Assesment of Lactulose vs Lactobacillus Acidophilus Effect in CKD Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman abobakr mokhtar, principal investigator, Assiut University
Other Study IDs: lactulose in CKD patients .
Record Dates: First submitted 2023-06-15; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: CKD
MeSH Terms: interventions — Lactulose; Lacteol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Lactulose — lactulose and lactobacillus acidophilus on ckd patients
  Other Names: lactobacillus acidophilus

SUMMARY:
Assessment for usage of laxatives and probiotics ,and its role in improving uremic parameters of CKD as GFR, UREA ,CREATININE, CLINICAL and UREMIC assessment (lower limb edema ,UOP,base of chest ,vomiting ,dyspnea,blood pressure measurement)

DETAILED DESCRIPTION:
with advanced CKD stages ,also have been linked to the high prevalence of constipation in CKD,Lactulose is a synthetic disaccharide.Lactulose is poorly absorbed from the gastrointestinal tract remains virtually unchanged and is then fermented by gut microbiota that increase osmotic effects and intraluminal gas formation . lactulose reduces the nitrogen products and urea, creatinine, uric acid, and b2- microglobulin levels. Lactulose also suppress tubulointerstitial fibrosis in a rat model of a kidney disease study . Lactulose modifies the gut microbiota, increasing the abundance of Bifidobacteria and Lactobacilli after 8 weeks of 30 ml lactulose syrup thrice daily, and ameliorates CKD progression by suppressing uremic toxin production .probiotics include vast array of products with living organisms whose purpose is to improve intestinal microbial balance and produce beneficial effect on ones health .probiotics is an alternative therapy for patients with CKD

ELIGIBILITY:
Inclusion Criteria:

* CKD stages 3,4,5 with non-dialysis receiving a diagnosis of constipation
* DM nephropathy

Exclusion Criteria:

* IBS (ulcerative colitis -crohns)
* HCV ,HBV ,
* autoimmune patients,
* malignancy pt
* cirrhotic patients
* haemodialysis patients
* cardiovascular patients
* abdominal surgery,
* gut obstruction,
* pregnancy,
* patients with ESRD on dialysis,
* history of lactulose allergy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 1. group A (50 PT DM and Non DM CKD Stage 3,4,5 not ON dialysis and receive lactulose 30 ml per day divided in 3 doses
  2. -group B (50 patients DM and Non DM CKD stage 3.4,5 not on dialysis and receive lactobacillus acidophilus one tab twice daily
  3. Group C control group (50 PT DM and Non DM CKD stage 3,4,5 not on dialysis and receive neither lactulose ,nor lactobacillus acidophilus .
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Assessment for usage of laxatives and probiotics ,and its role in improving uremic parameters in CKD patients and compare between both. | 1 year
  Assessment for usage of laxatives and probiotics ,and its role in improving uremic parameters in CKD patients and compare between both.

REFERENCES:
- [Background] Tayebi Khosroshahi H, Habibzadeh A, Khoshbaten M, Rahbari B, Chaichi P, Badiee AH. Lactulose for reduction of nitrogen products in patients with chronic kidney disease. Iran J Kidney Dis. 2014 Sep;8(5):377-81. PMID 25194404
- [Background] Tayebi-Khosroshahi H, Habibzadeh A, Niknafs B, Ghotaslou R, Yeganeh Sefidan F, Ghojazadeh M, Moghaddaszadeh M, Parkhide S. The effect of lactulose supplementation on fecal microflora of patients with chronic kidney disease; a randomized clinical trial. J Renal Inj Prev. 2016 Jul 29;5(3):162-7. doi: 10.15171/jrip.2016.34. eCollection 2016. PMID 27689115